CLINICAL TRIAL: NCT03671070
Title: Role of Low Dose Epinephrine Boluses For Acute Hypotension in The Pediatrics ICU
Brief Title: Role of Low Dose Epinephrine Boluses In Acute Hypotension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed E Eldaly, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RLDEBAH
Record Dates: First submitted 2018-09-07; First posted 2018-09-14 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Hypotension and Shock
MeSH Terms: conditions — Hypotension; Shock | interventions — Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose Epinephrine boluses (Active Comparator): Patients suffering from acute hypo-tension will receive low dose IV epinephrine boluses ≤ 5 μg/kg/dose, 3 doses, within 3 hours
  Interventions: Drug: Epinephrine
- Traditional management of shock (Placebo Comparator): Patients suffering from acute hypo-tension will be managed according to Traditional algorithm of Hypotension
  Interventions: Drug: Traditional management of shock

INTERVENTIONS:
Drug: Epinephrine — IV Low dose Boluses
  Other Names: Adrenaline
  Arms: Low dose Epinephrine boluses
Drug: Traditional management of shock — 1. Initial resuscitation: Push boluses of 20 cc/kg isotonic saline or colloid up to and over 60 cc/kg until perfusion improves or unless rales or hepatomegaly develop
  2. Fluid refractory shock: Begin inotrope IV/IO. Use atropine/ketamine IV/IO/IM to obtain central access and airway if needed. Reverse cold shock by titrating central dopamine or, if resistant, titrate central epinephrine. Reverse warm shock by titrating central norepinephrine.
  3. Catecholamine resistant shock: Begin hydrocortisone if at risk for absolute adrenal insufficiency.
  Other Names: Traditional management of hypotension
  Arms: Traditional management of shock

SUMMARY:
The Study evaluates the role of low dose epinephrine boluses in management of acute hypo-tension VS The Traditional management of acute hypo-tension.

Half of the participants suffering from acute hypo-tension will receive low dose epinephrine boluses (≤ 5 µg/kg/dose) and the other half will receive traditional management of shock

DETAILED DESCRIPTION:
Epinephrine, due to its alpha-1 and beta-adrenergic effects, is considered an important part of the management of children with hypo-tension. Epinephrine is typically used as a continuous infusion (0.02-0.5 μg/kg/min) for severe sustained hypo-tension and as a bolus (0.01 mg/kg, maximum dose = 1 mg) for bradycardia, asystole, or pulse-less arrest. There are, however, clinical conditions that may benefit from smaller doses of bolus epinephrine. For example, brief periods of hypo-tension during medical procedures, intermittent hemodynamic instability, and augmentation of low blood pressure in a pre-arrest condition. While a resuscitation (or code) dose of epinephrine would be inappropriate (as it would cause an unacceptable large increase in blood pressure and heart rate [HR]), a smaller dose may be particularly useful.

Low-dose bolus vasopressors have been used for decades by anaesthesiologists to prevent post-re-perfusion injury after solid organ transplant, control cerebral oxygenation during anaesthesia and manage acute hypo-tension during spinal surgery. Recently, use of bolus dose phenyl-ephrine has been described in the emergency department setting to augment blood pressure during periods of hypo-tension surrounding intubation. Finally, free open access medical publications have provided some insight into using bolus dose pressors for acute hypotensive episodes in adults. However, there is few published data describing the use of low-dose vasopressor boluses in children.

ELIGIBILITY:
Inclusion Criteria:

* Patients experiencing acute hypotensive episodes whether brief or during or after medical or surgical procedures

Exclusion Criteria:

* Patients experiencing acute hypotensive episodes in arrest or pre-arrest situations

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
change of mean value of blood Pressure both systolic and diastolic according to age group | within 1 Hours after injection
  Assessment of patients' blood Pressure (both systolic and diastolic) will be at at the onset of acute hypo-tension and after every bolus of low dose epinephrine and pressure will be reassessed after 20 minutes from each bolus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reiter PD, Roth J, Wathen B, LaVelle J, Ridall LA. Low-Dose Epinephrine Boluses for Acute Hypotension in the PICU. Pediatr Crit Care Med. 2018 Apr;19(4):281-286. doi: 10.1097/PCC.0000000000001448. PMID 29319635